CLINICAL TRIAL: NCT00750139
Title: A Phase 3 Double-Blind, Randomized, Placebo-Controlled, Multicenter, Parallel Group Evaluation of the Efficacy and Safety of NAFT-500 in Subjects With Tinea Pedis
Brief Title: Multicenter Study of the Safety and Efficacy of NAFT-500 in Tinea Pedis
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Merz North America, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: MUS 90200-0736/1
Record Dates: First submitted 2008-09-08; First posted 2008-09-10 (Estimated); Results first posted 2013-01-29 (Estimated); Last update posted 2013-04-26 (Estimated); Status verified 2013-04

CONDITIONS: Tinea Pedis; Athlete's Foot
Keywords: Tinea Pedis; Athlete's foot
MeSH Terms: conditions — Tinea Pedis

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (4):
- 1 (Experimental): Naftin 2% cream applied daily for 2 weeks
  Interventions: Drug: NAFT-500
- 2 (Placebo Comparator): Placebo cream applied daily for two weeks
  Interventions: Drug: Placebo 2-weeks
- 3 (Active Comparator): Active comparator applied daily for 4 weeks
  Interventions: Drug: Naftin 1%
- 4 (Placebo Comparator): placebo cream applied daily for 4 weeks
  Interventions: Drug: Placebo 4-weeks

INTERVENTIONS:
Drug: NAFT-500 — topical cream 1 application every day up to 4 weeks weeks
  Arms: 1
Drug: Placebo 2-weeks — placebo cream 1 application every day for up to 4 weeks
  Arms: 2
Drug: Naftin 1% — topical allylamine cream applied once a day for up to 4 weeks
  Arms: 3
Drug: Placebo 4-weeks — topical placebo cream applied once a day for up to 4 weeks
  Arms: 4

SUMMARY:
A research study to compare the safety and effectiveness of an investigational medication called NAFT-500 to placebo, when used in subjects with tinea pedis (athlete's foot).

DETAILED DESCRIPTION:
To evaluate the efficacy and safety of NAFT-500 compared to placebo in the treatment of subjects with potassium hydroxide (KOH) and culture positive symptomatic tinea pedis.

ELIGIBILITY:
Inclusion Criteria:

1. Review and sign a statement of Informed Consent and HIPAA authorization.
2. For minors (less than 18 years), the parent/legal guardian must complete the informed consent process AND the subject must complete the assent process and sign the appropriate form (if age appropriate).
3. Males or non-pregnant females ≥12 years of age, of any race or sex. Females of childbearing potential must have a negative urine pregnancy test.
4. Presence of tinea pedis on one or both feet characterized by clinical evidence of a tinea infection (at least moderate erythema, moderate scaling, and mild pruritus)based on signs and symptoms.
5. KOH positive and culture positive baseline skin scrapings obtained from the site most severely affected or a representative site of the overall severity.
6. Subjects must be in good health and free from any clinically significant disease that might interfere with the study evaluations.
7. Subject must be able to understand the requirements of the study and willing to comply with the study requirements.

Exclusion Criteria:

1. A life-threatening condition (ex. autoimmune deficiency syndrome, cancer, unstable angina, or myocardial infarction) within the last 6 months.
2. Subjects with abnormal findings - physical or laboratory - that are considered by the investigator to be clinically important and indicative of conditions that might complicate interpretation of study results.
3. Subjects with a known hypersensitivity to study medications or their components.
4. Subjects who have a recent history or who are currently known to abuse alcohol or drugs.
5. Uncontrolled diabetes mellitus.
6. Hemodialysis or chronic ambulatory peritoneal dialysis therapy.
7. Current diagnosis of immunocompromising conditions.
8. Foot psoriasis, corns and/or callus involving any web spaces, atopic or contact dermatitis.
9. Severe dermatophytoses, onychomycosis (on the evaluated foot), mucocutaneous candidiasis, or bacterial skin infection.
10. Extremely severe tinea pedis (incapacitating).
11. Female subject who is pregnant or lactating, who is not using or does not agree to use an acceptable form of contraception during the study, or who intends to become pregnant during the study (females who are surgically sterilized or post menopausal for at least 2 years are not considered to be of childbearing potential).For the purposes of this study, acceptable forms of birth control include: oral contraceptives, contraceptive patches/implants, double barrier methods (e.g., use of condom and spermicide), IUD, and abstinence with second acceptable method should subject become sexually active.
12. Subjects using the following medications:

    * Topical anti-fungal therapy, foot/shoe powders, or topical corticosteroids applied to the feet within 14 days prior to randomization. Topical terbinafine, butenafine,and naftifine within 30 days prior to randomization
    * Oral anti-fungal therapies 3 months (8 months for oral terbinafine) prior to randomization
    * Systemic antibiotic or corticosteroid treatment within 30 days of randomization
    * Any other significant treatments, except hormonal contraception and multivitamin, at the discretion of the investigator that would interfere with study treatment.
    * Investigational drug within 30 days of randomization

Min Age: 12 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 707 (Actual)
Dates: Start 2008-08; Primary Completion 2009-08 (Actual); Study Completion 2009-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Lawrence Parish, MD, Principal Investigator — Paddington Testing Company
Locations (17):
- United States (17):
  - Radiant Research, Birmingham, Alabama
  - Dr. Felix Sigal, Los Angeles, California
  - University of California San Francisco, Dept of Dermatology, San Francisco, California
  - FXM Research, Miami, Florida
  - FXM Research, Miramar, Florida
  - Glazer Dermatology, Buffalo Grove, Illinois
  - Tulane University Health Services, New Orleans, Louisiana
  - Silverton Skin Institute, Grand Blanc, Michigan
  - Zoe Draelos, MD, High Point, North Carolina
  - Haber Dermatology, Euclid, Ohio
  - Oregon Dermatology and Research Center, Portland, Oregon
  - Paddington Testing Company, Philadelphia, Pennsylvania
  - Temple University School of Podiatric Medicine, Philadelphia, Pennsylvania
  - Coastal Carolina Research Center, Mt. Pleasant, South Carolina
  - J & S Studies, College Station, Texas
  - Research Across America, Dallas, Texas
  - Research Across America, Plano, Texas

REFERENCES:
- [Derived] Parish LC, Parish JL, Routh HB, Fleischer AB Jr, Avakian EV, Plaum S, Hardas B. A randomized, double-blind, vehicle-controlled efficacy and safety study of naftifine 2% cream in the treatment of tinea pedis. J Drugs Dermatol. 2011 Nov;10(11):1282-8. PMID 22052309

RESULTS

PARTICIPANT FLOW:
Groups:
- NAFT-500: Naftin 2% Cream applied daily for 2 weeks
- Placebo 2-wks: Placebo applied daily for 2-weeks
- Naftin 1%: Naftin 1% active comparator applied daily for 4 weeks
- Placebo 4-wks: Placebo cream applied daily for 4 weeks
Period: Overall Study
Arm/Group | NAFT-500 | Placebo 2-wks | Naftin 1% | Placebo 4-wks
Started | 234 | 118 | 236 | 119
Completed | 145 | 59 | 135 | 73
Not Completed | 89 | 59 | 101 | 46
Not completed — Adverse Event | 1 | 2 | 0 | 1
Not completed — Lost to Follow-up | 17 | 12 | 15 | 6
Not completed — Withdrawal by Subject | 3 | 2 | 6 | 2
Not completed — Physician Decision | 1 | 1 | 0 | 0
Not completed — Non-compliance | 1 | 0 | 1 | 3
Not completed — Termination by sponsor | 4 | 0 | 0 | 1
Not completed — Non-specific | 62 | 42 | 79 | 33

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | NAFT-500 | Placebo 2-wks | Naftin 1% | Placebo 4-wks | Total
Number analyzed (Participants) | 234 | 118 | 236 | 119 | 707
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 2 | 1 | 14 | 6 | 23
  Between 18 and 65 years | 220 | 115 | 212 | 111 | 658
  >=65 years | 12 | 2 | 10 | 2 | 26
Age Continuous [Mean (Standard Deviation); unit: years] | 42.7 (13.03) | 41.0 (12.91) | 41.4 (14.08) | 41.4 (14.00) | 41.7 (13.52)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 63 | 38 | 71 | 33 | 205
  Male | 171 | 80 | 165 | 86 | 502
Region of Enrollment [Number; unit: participants]
  United States | 234 | 118 | 236 | 119 | 707

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Subjects With Complete Cure at Week 6.
Description: The first primary efficacy variable was the percentage of subjects in the NAFT-500 Cream, 2% or 2-week placebo groups with complete cure at Week 6.
  The second primary efficacy variable was the percentage of subjects in the Naftin 1% Cream or 4-week placebo groups with complete cure at Week 6.
  Complete cure was defined as negative mycology results from the central laboratory (dermatophyte culture and KOH) and absence of erythema, scaling, and pruritus that were evaluated using a 4 point severity scale.
Time Frame: Week 6
Population: This is based on the Full Analysis Set (FAS). The FAS is the subset of all subjects in the Safety Evaluation Set (SES) with a positive culture at baseline for whom the primary efficacy variable is available. This is a modified intent to treat (MITT) principle because the culture results will not be available before the start of treatment.
Measure: Number; unit: percentage of subjects with complete cur
Groups:
- Placebo 2-weeks: Placebo Control cream applied daily for 2-weeks
- Placebo 4-wks: Placebo control cream applied daily for 4 weeks
Arm/Group | NAFT-500 | Placebo 2-weeks | Naftin 1% | Placebo 4-wks
Number analyzed (Participants) | 147 | 70 | 143 | 65
percentage of subjects with complete cur | 17.7 | 7.1 | 16.1 | 3.1
Statistical Analysis 1: Comparison: NAFT-500 vs Placebo 2-weeks; The first primary efficacy hypotheses tests are: H01: p1 ≤ p01 vs. H1: p1 > p01 where p01 and p1 denote the proportions of complete cure in the placebo 2wks and NAFT-500 groups, respectively; Test type: Superiority or Other; p = 0.010, Cochran-Mantel-Haenszel — The first primary efficacy analyses will use the Cochran-Mantel-Haenszel (CMH) test after stratification by pooled clinical site. The test will be conducted with the FAS at a one-sided level of significance of α = 0.025
Statistical Analysis 2: Comparison: Naftin 1% vs Placebo 4-wks; The second primary efficacy hypotheses tests are: H02: p2 ≤ P02 vs. H2: P2 > p02 where p02 and p2 are denote proportions of complete cure in the placebo 4wks and Naftin 1% groups, respectively; Test type: Superiority or Other; p = 0.001, Cochran-Mantel-Haenszel — The second primary efficacy analyses will use the Cochran-Mantel-Haenszel (CMH) test after stratification by pooled clinical site. The test will be conducted with the FAS at a one-sided level of significance of α = 0.025

2. Secondary Outcome: Percentage of Subjects With Mycological Cure and Percentage of Subjects With Treatment Effectiveness at Week 6
Description: Mycological Cure was defined as negative KOH result and negative dermatophyte culture at Week 6. Treatment Effectiveness was defined as negative KOH, negative culture, and Scaling, Erythema, and Pruritus grades of 0 or 1 at Week 6.
Time Frame: Week 6
Population: This was the Full Analysis Set (FAS) comprising of subjects in the Safety Evaluation Set (SES) with a positive culture at baseline for whom the primary efficacy variable was available. This was a Modified Intent to Treat (MITT) principle because the culture results were not available at the start of treatment.
Measure: Number; unit: percentage of Subjects
Arm/Group | NAFT-500 | Placebo 2-wks | Naftin 1% | Placebo 4-wks
Number analyzed (Participants) | 147 | 70 | 143 | 65
percentage of Subjects
  Mycological Cure (MC) | 67.3 | 21.4 | 71.3 | 21.5
  Treatment Effectiveness (TE) | 56.5 | 20.0 | 58.7 | 13.8

ADVERSE EVENTS:
Arm/Group | NAFT-500 | Placebo 2-wks | Naftin 1% | Placebo 4-wks
Serious Adverse Events (participants affected / at risk) | 0/234 | 0/118 | 1/236 | 0/119
Other Adverse Events (participants affected / at risk) | 38/234 | 22/118 | 31/236 | 26/119
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | NAFT-500 (N=234) | Placebo 2-wks (N=118) | Naftin 1% (N=236) | Placebo 4-wks (N=119)
Influenza (Infections and infestations) | 0 | 0 | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | NAFT-500 (N=234) | Placebo 2-wks (N=118) | Naftin 1% (N=236) | Placebo 4-wks (N=119)
Headache (Nervous system disorders) | 10 | 4 | 9 | 3
Nasopharyngitis (Infections and infestations) | 3 | 2 | 5 | 4
Application Site Irritation (General disorders) | 4 | 3 | 4 | 5
Application Site Pruritus (General disorders) | 7 | 4 | 1 | 3
Pain (General disorders) | 4 | 3 | 4 | 5
Application Site Dryness (General disorders) | 4 | 2 | 1 | 0
Blood Creatinine Increased (Investigations) | 1 | 2 | 2 | 1
Alanine Aminotransferase Increased (Investigations) | 1 | 0 | 2 | 2
Blood Glucose Increased (Investigations) | 1 | 2 | 0 | 1
Protein Urine Present (Investigations) | 1 | 2 | 0 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 2 | 2 | 3 | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Institution and Principal Investigator agree not to individually publish the results of the Study. Institution and Principal Investigator may, however, upon written notice to Merz participate in a joint, multicenter publication of the Study results with other investigators and/or institutions, provided that the manuscript or abstract is first reviewed by Merz.